CLINICAL TRIAL: NCT04725929
Title: Vaginal Progesterone as Prophylactic Against a Second Attack of Antepartum.Haemorrhage in Pregnant Women Diagnosed as Placenta Previa
Brief Title: Vaginal Progesterone Against a Second Attack of Antepartum Haemorrhage in Placenta Previa Women
Status: Completed | Type: Observational
Sponsor: Nourhan Ashraf ElSherbiny (Other)
Responsible Party: Sponsor-Investigator, Nourhan Ashraf ElSherbiny, The principal.investigator, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: Placenta Previa
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Placenta praevia is associated with an increased risk of preterm delivery (PTD) especially if associated with bleeding and uterine contractions .

In this study we will determine the effect of Progesterone in preventing a second attack of antepartum haemorrhage in pregnant women diagnosed with placenta previa

DETAILED DESCRIPTION:
Placenta previa is a problem of pregnancy in which the placenta grows in the lowest part of the womb (uterus) and covers all or part of the opening to the cervix .

The prevalence of placenta previa has been recently estimated to be approximately 0.5% of all pregnancies, and this increase correlates to the elevated cesarean section rate .

Placenta previa is a major cause of maternal morbidity and mortality because of the associated massive antepartum and intrapartum hemorrhage .

Moreover, placenta previa is associated with preterm delivery, with the neonatal mortality increasing threefold as a result of prematurity. Although placenta previa is associated with antepartum hemorrhage, massive hemorrhage necessitating preterm cesarean section is not observed in all women with the condition .

The term placenta praevia should be used when the placenta lies directly over the internal os. For pregnancies at more than 16 weeks of gestation the term low-lying placenta should be used when the placental edge is less than 20 mm from the internal os on transabdominal or transvaginal scanning (TVS) .

If the placenta is thought to be low lying (less than 20 mm from the internal os) or praevia (covering the os) at the routine fetal anomaly scan, a follow-up ultrasound examination including a TVS is recommended at 32 weeks of gestation to diagnose persistent low-lying placenta and/or placenta praevia The ability to predict severe antepartum hemorrhage and emergency cesarean section is critical in the management of placenta previa To date, no consensus exists on the preterm delivery risk of different types and locations of placenta previa (Fan et al., 2017). Only a few reports have focused on the maternal and perinatal outcomes of different types of placenta previa .

Furthermore, the effect of anterior/posterior placental position on preterm delivery is unknown, although increased perinatal risks, including placenta previa, excessive intraoperative blood loss, hysterectomy, and neonatal anemia, have been reported to be associated with anterior placenta previa .

The symptomatic placenta previa are being treated with tocolytic agents. The progesterone is necessary for the preservation of pregnancy and aids in the extension of pregnancy The progesterone, also known as pregn-4-ene-3, 20-dione is an endogenous steroid and involved in the menstrual cycle, pregnancy, and embryogenesis of humans . It is included in a steroid hormone group known as progestogens.

The progesterone is also a key metabolic intermediate in the making of other endogenous steroids such as the sex hormones and the corticosteroids . They show a vital part in brain function as a neurosteroid.

Reduction of the rate of long-term morbidity requires delayed delivery which facilitates the maturity of vital organs. Though the thorough mechanism of action is not known but proposed mechanisms were: (a) It acts principally through creating uterine inertness and upholds cervical length. It has immunosuppressive activity and stops consequence of oxytocin on myometrium. (b) It is a powerful inhibitor of gap junctions between myometrial cells. (c) Local fluctuations in progesterone or estrogen or progesterone ratio. (d) Suppression of calcium-calmodulinmyosin light chain kinase system, decreasing calcium flux and shifting the resting potential of smooth muscle are the root of progesterone action

72. AIM/ OBJECTIVES This study aims to determine the effect of vaginal progesterone in preventing a second attack of antepartum haemorrhage in pregnant women diagnosed with placenta previa.

Research Question:

Does vaginal progesterone prevent a second attack of antepartum haemorrhage in pregnant women diagnosed with placenta previa?

Research hypothesis:

Vaginal progesterone prevents the second attack of antepartum haemorrhage in pregnant women diagnosed with placenta previa.

3. METHODOLOGY: Patients and Methods/ Subjects and Methods/ Material and Methods

* Type of Study:double blinded randomised controlled clinical trial.
* Study Setting: Ain Shams university, Maternity hospital, Faculty of medicine-Ain Shams university.
* Study Period: January 2021-july 2021 or until completing the required cases.
* Study Population:

Pregnant women diagnosed with placenta praevia. • Ethical considerations: The study will be approved from the Ethical Committee of the Department of Obstetrics and Gynecology, Faculty of Medicine, Ain Shams University.

Informed written consents will be taken from all women before recruitment in the study, and after extensive explanation and clear discussion of risks and benefits.

This study will be conducted on female patients at Ain Shams maternity hospital. The participants included in the study will meet the following included and excluded criteria.

• Selection criteria for cases:

Inclusion Criteria:

* Women diagnosed as placenta previa.
* Women aged 20-40 years, who were pregnant in a single foetus
* Gestational age ranging between 24 and 34 weeks
* Patient had attack of Antepartum Haemorrhage or history of Antepartum Haemorrhage

Exclusion Criteria:

Patients with:

* History of previous PTD
* Polyhydramnios
* Severe attack of bleeding requiring an immediate intervention
* Intrauterine foetal death

  * Sampling method: Convenience sampling
  * Sample Size: Using PASS 11 program for sample size calculation, confidence level 90%, margin error +/- 0.1, and by reviewing previous studies (Singh and Jain, 2015), showed the rates of recurrent bleeding among patients taking progesterone versus patients taking placebo were (77.5%vs 87.5% respectively); based on that, the required sample size will be 80 patients in each group to be sufficient to detect the difference between groups.
  * Patients and Methods (Methodology):

This study included two groups:

* Group I, vaginal Progesterone (Vaginal progesterone "prontogest 400 MG") Once Daily starting from 24 to 34 weeks of gestation or rectal progesterone if the patient fears of taking vaginal or still have bleeding,
* Group II, included placenta praevia patients receiving a placebo

Randomisation:

Randomisation will be conducted using a computer-generated table of random numbers with allocation concealment. Once allocation has been done, it will not be changed.

Follow up schedule:

The women with placenta previa who have attack of antepartum haemorrhage or history or attack will be admitted in the hospital and kept under observation for 48 hours, and will be encouraged to go home and continue follow up at our outpatient Obstetric Clinic every 1-2 weeks (according to patients' compliance).

All placenta praevia women with severe attack of antepartum haemorrhage will be encouraged to remain in hospital until bleeding stops or up to delivery.

They will receive prophylactic corticosteroids. Parenteral iron supplementation will be needed for optimal correction of anaemia in both groups (mean haemoglobin [Hb] level was 9 g/dL).

During follow-up visits, women will carefully be asked about abdominal pain, number and amount of vaginal bleeding attacks.

Unscheduled ultrasound examinations ± cardiotocography (CTG) will be done for foetal-maternal indications as a heavy attack of bleeding, decreased foetal movement, suspected preterm premature rupture of the membranes (PROM) or PTL.

Patients with features suggestive of placenta previa spectrum will carefully be examined and followed by an expert sonographer using 2D grey scale imaging and colour Doppler imaging, according to the guidelines of the European Working Group on Abnormally Invasive Placenta used for the prenatal diagnosis of placenta previa.

you follow the Royal College of Obstetricians' and Gynaecologists' guidelines as regards the time of elective delivery in placenta praevia women, so patients were delivered when completed 37 weeks of gestation .

Our hospital protocol for placenta praevia delivery recommends delivery at 37-38 weeks because of limited neonatal services in our country or earlier if the women developed another severe attack of antepartum haemorrhage, developed contractions.

ELIGIBILITY:
Inclusion Criteria:

* o Women diagnosed as placenta previa.

  * Women aged 20-40 years, who were pregnant in a single foetus
  * Gestational age ranging between 24 and 34 weeks
  * Patient had attack of Antepartum Haemorrhage or history of Antepartum Haemorrhage

Exclusion Criteria:

* o History of previous PTD

  * Polyhydramnios
  * Severe attack of bleeding requiring an immediate intervention
  * Intrauterine foetal death

Ages: 24 Weeks to 34 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: * Group I, vaginal Progesterone (Vaginal progesterone "prontogest 400 MG") Once Daily starting from 24 to 34 weeks of gestation or rectal progesterone if the patient fears of taking vaginal or still have bleeding,
  * Group II, included placenta praevia patients receivinv placebo
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
patient with past history of antepartum haemorrhage will not have a secondary attack | 2 weeks
  decrease the bleeding

SECONDARY OUTCOMES:
duration between first and secondary attack | 2 week
  time between primary and secondary attack

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ghaleb, MD, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt